CLINICAL TRIAL: NCT05114551
Title: ICU Predictive Score of WEaning Success in Patients At Risk of Extubation Failure
Acronym: I-SWEAR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: I -Swear (RNI 2021 AUDARD)
Record Dates: First submitted 2021-10-29; First posted 2021-11-10 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Mechanical Ventilator Weaning; Predictive Value of Tests; Ventilator Weaning; Airway Extubation; Care Unit, Intensive; Critical Care; Area Under Curve; Sensitivity and Specificity; Logistic Models; Prospective Studies; Echocardiography, Transthoracic; Ultrasonography; Biomarkers / Blood
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Observational study in two medical-surgical intensive care units of the Clermont-Ferrand University Hospital to develop a composite score for prediction of 72h-extubation failure in patients at risk of extubation failure.

DETAILED DESCRIPTION:
In our intensive care units, when a patient does not have risk factors for extubation failure, SBT (Spontaneous Breathing Trial) in PSV (Pressure Support Ventilation) is usually performed first as recommended. If patient fails the first SBT in PSV or extubation, weaning is considered difficult (WIND study group AJRCCM 2017). In this case, the service protocol provides a T-piece SBT for the following SBT. In addition, this same protocol proposes to perform T-piece SBT from the first weaning event in patients with risk factors for WiPO (Weaning-induced Pulmonary Oedema), defined as obesity (BMI >30 kg/m2), COPD (Chronic Obstructive Pulmonary Disease) (suspected or known), or heart disease (structural [hypertrophic, dilated, valvular], functional [diastolic or systolic dysfunction], ischemic, or dysrhythmic).

Our study population concerns patients for whom a T-piece trial is performed according to the service protocol.

A patient is potentially includible in the study if he has been under mechanical ventilation for at least 48h and if he presents criteria of weanability with a planned T-piece SBT. As long as the inclusion and non-inclusion criteria are respected (see inclusion/non-inclusion criteria), clinical, biological and ultrasound data will be collected before and at the end of the ventilatory weaning test. If the patient fails the weaning test and/or is not extubated following the test, data from each new T-piece SBT will be collected within 7 days of inclusion.

The global management of the patient, before, during and after the inclusion of the patient in the study is the one usually practiced in our intensive care units, based on the national and international recommendations as well as the literature exposed in the protocol.

During the patient's stay in the ICU, data from the medical record will be collected (demographic, clinical, treatment, vital status,...). A follow-up at D7, D28 and D90 will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Invasive mechanical ventilation for at least 48 hours
* Criteria for ventilatory weaning are present
* T-piece spontaneous breathing trial planned
* Patients with a social security program

Exclusion Criteria:

* Patients already included in this study during the same stay in intensive care
* Resuscitation neuromyopathy defined by an MRC (Medical Research Council) score < 48/60
* Surgery planned within 72 hours
* Prolonged ventilatory weaning (>7 days after the first SBT)
* Patients with tracheostomy
* Patients with non-reintubation decision or terminal extubation
* Brain damaged patients
* Patients with ECMO/ECLS
* Tetraplegic or paraplegic patients with lesion level higher than T8
* Nasotracheal intubated patients
* Pregnant or breastfeeding women
* Refusal to participate in the study (refusal by patient or family member/trusted person).
* Patients under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients included in this study will be all the patients hospitalized in our 2 intensive care units, under mechanical ventilation for at least 48h, meeting the criteria of weanability and for whom a T-piece SBT will be planned.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-09-28 (Actual); Primary Completion 2023-09-28 (Estimated); Study Completion 2023-09-28 (Estimated)

PRIMARY OUTCOMES:
The primary outcome measure is extubation failure, defined as the need for reintubation within 72 hours of extubation. | 72 hours

SECONDARY OUTCOMES:
Mortality at day 7, 28 and 90 | 90 days
Length of stay in intensive care | 90 days
Number of days without mechanical ventilation from study inclusion to day 28 | 28 days
Time frame and reasons for reintubation in case of failed extubation. | 28 days
Use of non-invasive post-extubation ventilation | 7 days
Use of High Flow Nasal Oxygenation post-extubation | 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- CHU, Clermont-Ferrand, France